CLINICAL TRIAL: NCT00317005
Title: Randomized Clinical Trial of Folate Therapy/Placebo for Reduction of Homocysteine Serum Levels in Uremic Patients and Influence on Cardiovascular Mortality
Brief Title: Uremic Hyperhomocysteinemia -A Folate Trial for Possible Prevention of Cardiovascular Events
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UEL/CPG/Nefro/Hcy
Record Dates: First submitted 2006-04-18; First posted 2006-04-21 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2005-05

CONDITIONS: Uremia; Chronic Renal Failure; Hemodialysis; Hyperhomocysteinemia; Cardiovascular Disease
Keywords: hemodialysis; chronic uremia; hyperhomocysteinemia; folate
MeSH Terms: conditions — Uremia; Kidney Failure, Chronic; Hyperhomocysteinemia; Cardiovascular Diseases

INTERVENTIONS:
Drug: folate treatment

SUMMARY:
Homocysteine recently gained access to the category of risk factor for the development of atherosclerotic cardiovascular disease in the general population. Chronic renal failure patients, even before being introduced to dialysis therapy have almost universal elevation of serum homocysteine; when on dialysis their mortality is above 50% related to cardiovascular disease that we might now speculate, with a contribution of potentially toxic levels of the aminoacid homocysteine.

DETAILED DESCRIPTION:
We conducted a double blind , randomized, placebo controlled trial, for two years, enroling, simultaneously, 186 end-stage kidney disease patients of any cause, older than 18 years of age, stable on hemodialysis, assigned to receive either oral folic acid 10 mg three times a week on post dialysis sessions, under nurse supervision or an identical appearing placebo for the entire lenght of the study, from april 2003 to march 2005.

The two groups had similar baseline clinical and laboratory characteristics. There was no loss of follow-up. At admission, homocysteine serum levels were above 13,9 umol/L in 96.7% (median 25.0, range 9.3-104.0)with only five cases in the normal levels; homocysteine remained elevated at 6, 12 and 24 months on those receiving placebo; folate treatment significantly decreased total homocysteine levels to a median value of 10.5 umol/L (2.8 - 20.3)which remained at this level for the entire study time (P<0.001); every one was alive and tested at six months, sixty eight were either transplanted(15)or died (53) from cardiovascular disease(seventeen in the folic acid group and twenty one in the placebo (P>0.05)or other causes(15), after being included in the study. Intima-media wall thickness blinded measured at the common carotid artery decreased from 1.94+-0,59 mm to 1.67+-0.38 (P<0.001) with folate therapy and became thicker, from 1.86+-0.41 to 2.11+-0.48 mm in the placebo group.

In conclusion, folate treatment for two years was not effective on modifying cardiovascular death and non fatal cardiovascular events of this sample population with chronic uremia; however, the ultrasonographic evaluation of the common carotid arteries intima-media wall thickness at entry and twenty four months later unequivocally showed a significant thickness decrease with supervised folate intake.

Earlier prescription of folic acid might benefit patients with chronic renal failure,preventing cardiovascular deterioration

ELIGIBILITY:
Inclusion Criteria:

* Patients stable on hemodialysis for 4 months or more
* Eighteen years of age or older

Exclusion Criteria:

* Potential kidney transplant from a living donor in the near future
* Severe cardiovascular disease
* Cancer and active inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186
Dates: Start 2003-04; Study Completion 2005-03

PRIMARY OUTCOMES:
Lowering of Homocysteine blood levels in uremia.
Prevention of cardiovascular events

SECONDARY OUTCOMES:
Reduction of carotid intima-media thickness

CONTACTS AND LOCATIONS:
Overall Officials: Altair J Mocelin, MD PHD, Study Director — Nephrology, University Hospital, State University of Londrina
Locations (2):
- Brazil (2):
  - Hospital Universitario regional do Note do Parana, Londrina, Paraná
  - University Hospital, State University of Londrina, Londrina, Paraná

REFERENCES:
- [Background] Brenner RM, Wrone EM. The epidemic of cardiovascular disease in end-stage renal disease. Curr Opin Nephrol Hypertens. 1999 May;8(3):365-9. doi: 10.1097/00041552-199905000-00015. No abstract available. PMID 10456270